CLINICAL TRIAL: NCT02274623
Title: Effect of CTAP101 Capsules on Serum Calcium, Plasma Intact Parathyroid Hormone and Vitamin D Metabolites in Patients With Advanced Breast or Prostate Carcinomas With Metastases to Bone and Receiving Ongoing Therapy With Denosumab or Zoledronic Acid
Brief Title: Effect of CTAP101 Capsules on Ca/iPTH in Advanced Breast/Prostate Cancer Patients Treated With Denosumab/Zoledronic Acid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CTAP101-CL-1017
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Breast Cancer; Prostate Cancer; Bone Neoplasms; Hypocalcemia; Hyperparathyroidism, Secondary
Keywords: Bone Neoplasms; Hypocalcemia; Hyperparathyroidism, Secondary
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Bone Neoplasms; Hypocalcemia; Hyperparathyroidism, Secondary | interventions — Calcifediol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CTAP101 Capsules (Experimental): CTAP101 Capsules daily
  Interventions: Drug: CTAP101 Capsules

INTERVENTIONS:
Drug: CTAP101 Capsules — escalating doses
  Other Names: calcifediol

SUMMARY:
This is an open-label exploratory study of CTAP101 Capsules in patients with bone metastases arising from either breast or prostate cancer, who are taking anti-resorptive therapy.

DETAILED DESCRIPTION:
This is a multi-center, open-label, repeat-dose study to evaluate the safety, efficacy, and tolerability of CTAP101 Capsules in subjects with bone metastases who are receiving ongoing therapy with denosumab or zoledronic acid. Following screening, approximately 12 eligible subjects with breast cancer and approximately 12 eligible subjects with prostate cancer, all of whom have metastases to bone and are undergoing treatment with anti-resorptive therapies, will receive CTAP101 Capsules at an initial daily oral dose of 30 μg (1 capsule) for 4 weeks. The daily dose may be increased in 30 μg (1 capsule) increments at 4-week intervals to a maximum of 300 μg or until serum calcium reaches >10.3 mg/dL for two consecutive visits (dose escalation phase) at which time the subject will suspend dosing until serum calcium is ≤10.0 mg/dL and will directly enter a 12-week maintenance phase, resuming treatment at a reduced daily dose, followed by a 2-week follow-up period. Subjects reaching the maximum dose without serum calcium reaching >10.3 mg/dL, will directly enter the 12-week maintenance phase, followed by a 2-week follow-up period. Serum markers for monitoring bone metabolism (including plasma iPTH, PTHrP, and serum free calcifediol), immune function and tumor burden will be measured during the treatment period. The FACT-BP Quality of Life Measurement in Patients with Bone Pain questionnaire will be used to explore the effect of the treatment, if any, on musculoskeletal pain. The genotype of vitamin D binding protein (DBP) will also be determined. Safety will be monitored through adverse events, serum and urine chemistries, hematology, and ECGs.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with bone metastases subsequent to breast (female subjects only) or prostate carcinoma, and will have received zoledronate or denosumab therapy for at least 3 months at the time of enrollment
* Be at least 18 years of age
* Have a life expectancy >12 months from the anticipated time of initiation of treatment
* Serum calcium <9.8 mg/dL
* Plasma iPTH ≥70 pg/mL if taking <1200 IU vitamin D
* Estimated glomerular filtration rate (GFR) >15 mL/min/1.73m2
* If taking more than 1000 mg/day of elemental calcium, must be willing and able to discontinue or reduce their calcium use and/or use non-calcium based therapies for the duration of the study
* Subjects receiving ≤2000 IU/day vitamin D (ergocalciferol or cholecalciferol) therapy must remain on a stable dose during the study. If taking more than 2000 IU/day of vitamin D (ergocalciferol or cholecalciferol), must be willing and able to reduce use to ≤2000 IU/day and remain on a stable dose for the duration of the study
* Is willing and able to comply with study instructions and commit to all clinic visits for the duration of the study
* Female subject of childbearing potential is neither pregnant nor lactating and must have a negative pregnancy test at the screen visit and a negative pregnancy test before dosing. All female subjects of childbearing potential and male subjects with female partners of childbearing potential must agree to use effective contraception (eg, implants, injectables, combined oral contraceptives, intrauterine device (IUD), sexual abstinence, vasectomy or vasectomized partner) for the duration of the study
* Has the ability to read and understand subject Informed Consent Form (ICF).

Exclusion Criteria:

* Spot urine Ca:Cr ratio >0.25 (>250 mg/g creatinine)
* Known previous or concomitant serious illness (other than advanced cancer with metastatic bone disease) or medical condition, such as, HIV, significant gastrointestinal disease, or cardiovascular event that in the opinion of the investigator may worsen and/or interfere with participation in the study
* History of neurological/psychiatric disorder, including psychotic disorder or dementia, or any other reason, which in the opinion of the investigator makes adherence to a treatment or follow-up schedule unlikely
* Known or suspected hypersensitivity to any of the constituents of the investigational product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2014-12; Primary Completion 2017-02-27 (Actual); Study Completion 2017-03-17 (Actual)

PRIMARY OUTCOMES:
Effect of repeated, escalating doses of CTAP101 on serum calcium and plasma iPTH levels | up to 52 weeks
Effect of repeated, escalating daily doses of CTAP101 on serum calcifediol | up to 52 weeks
Safety and tolerability of CTAP101 | up to 52 weeks
  Measured by the number of participants with treatment related adverse events and abnormal physical examinations, vital signs, clinical laboratory tests (hematology, coagulation, and clinical chemistry, urine calcium, albumin and creatinine), and 12-lead ECG.

SECONDARY OUTCOMES:
Effect of repeated, escalating daily doses of CTAP101 on vitamin d metabolites | up to 52 weeks
Effect of repeated, escalating doses of CTAP101 on serum phosphorus and spot urine calcium:creatinine ratio | up to 52 weeks

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Coast Hematology-Oncology Associates, Long Beach, California
  - Mount Sinai Medical Center, Comprehensive Cancer Center, Miami, Florida
  - Research by Design LLC, Evergreen Park, Illinois
  - Roswell Park Cancer Institute, Buffalo, New York
  - University of Cincinnati Cancer Institute, Cincinnati, Ohio
  - Inova Dwight and Martha Schar Cancer Center, Fairfax, Virginia